CLINICAL TRIAL: NCT06835426
Title: High-resolution PET-CT Specimen Imaging for the Perioperative Visualization of Resection Margins: an Exploratory Pilot Study
Brief Title: High-resolution PET-CT Specimen Imaging for the Perioperative Visualization of Resection Margins
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Tessa Van Oostveldt, Principal Investigator, Algemeen Ziekenhuis Maria Middelares
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MMS.2022.048; B0172022000009 (Registry Identifier: BUN number (Raadgevend Comité voor Bio-ethiek))
Record Dates: First submitted 2024-12-13; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Breast Carcinoma; Prostate Cancer Surgery; Thyroid Cancer; Parathyroid Adenomas; Skin Cancer; Genitourinary Cancer; Head and Neck Cancer; Hepatobiliary Cancers; Metabolic Abnormality; Neuro Endocrine Tumours; Brain Tumours; Gastro Intestinal Cancer; Thoracoscopic Surgery
Keywords: resective surgery; perioperative high-resolution PET-CT specimen imaging; breast cancer; Prostate cancer; thyroid cancer; parathyroid cancer; head and neck cancer; neuro-endocrine malignancies; genitourinary malignacies; thoracovascular malignancies
MeSH Terms: conditions — Breast Neoplasms; Thyroid Neoplasms; Parathyroid Neoplasms; Skin Neoplasms; Urogenital Neoplasms; Head and Neck Neoplasms; Brain Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The rationale of this pilot study is to obtain scientific knowledge on the clinical usefulness of perioperative high-resolution PET-CT specimen imaging in different clinical indications and to document the radiation safety of perioperative high-resolution PET-CT specimen imaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): This is a single-arm interventional pilot study. Patients eligable for this study who signed the Informed consent will be included and will follow the interventions as described.
  Interventions: Other: Single intravenous injection of the radiotracer; Diagnostic Test: Imaging resected specimen using the high-resolution PET-CT specimen imager

INTERVENTIONS:
Other: Single intravenous injection of the radiotracer — * only in case of 18F-FDG as PET-tracer: blood glucose level is measured;
  * single intravenous injection of the radiotracer between 30 minutes and 5 hours (ideally between 60 and 90 minutes) before the specimen is imaged. The type and dose of radiotracer depends on the patient group:
    * breast cancer group: 0.8 MBq/kg of 18F-FDG
    * prostate cancer group: 1 MBq/kg 18F-PSMA
    * thyroid cancer group: 1 MBq/kg of 18F-FDG
    * parathyroid adenoma group: 1 MBq/kg of 18F-Choline
    * head & neck cancer group: 1 MBq/kg of 18F-FDG
    * skin cancer group: 4 MBq/kg of 18F-FDG
    * primary and secondary hepatobiliary tumors group: 1 MBq/kg of 18F-FDG
    * genitourinary malignancies group: 1 MBq/kg of 18F-FDG
    * metabolic active lesions undergoing biopsy: 1 MBq/kg of 18F-FDG
    * Neuro-endocrine malignancies group: 1 MBq/kg of 18F-FDG
    * Brain tumor group: 1 MBq/kg of 18F-FDG, 18F-Choline or 18F
    * Gastrointestinal group: 1 MBq/kg of 18F-FDG
    * Thoracovascular group: 1MBq/kg of 18F-FDG
Diagnostic Test: Imaging resected specimen using the high-resolution PET-CT specimen imager — * the resected specimen is imaged in the operation theatre using the high-resolution PET-CT specimen imager (XEOS Aura; XEOS Medical, Ghent, Belgium); in principle no treatment decisions will be taken based on the images acquired by the specimen imager; however a decision to extend the resection can be taken at the discretion of the surgeon if there is clinical suspicion of a positive resection margin;
  * additional resected tissue (e.g. lymph nodes, cavity shaves etc) could also be imaged by the high-resolution PET-CT specimen imager; no treatment decisions will be taken based on the images acquired by the specimen imager;

SUMMARY:
These are patients in whom a benign or malignant tumor was recorded requiring surgery. During that surgery, the surgeon will cut away the tumor as part of the treatment of the disease. In this process, it is important that the tumor is removed correctly and completely. To verify that the correct tissue was completely removed, the tissue is examined microscopically. However, a microscopic analysis takes a relatively long time and the result is not known until a few days after the surgery is completed. If that microscopic analysis should eventually reveal that the tumor was not completely removed, additional treatment is usually necessary. An assessment of the excised tissue during surgery would allow additional tissue to be excised in the same operation if necessary. Thus, in this way, additional treatments can also be avoided. This could lead to shorter treatment time and less emotional strain for the patient, as well as lower costs. To date, however, there are no effective techniques to do this.

PositronEmissionTomography (PET) imaging can be used to image the tumor that needs to be excised. To do this, a tracer must be administered through the blood before the operation. This tracer is a slightly radioactive substance that can be detected by the PET camera even at low concentrations. This technique is already routinely used in the hospital to detect cancer or inflammatory tissue in the body. During this study, however, it's not the intention to look at the tumor while it is still in the patient's body, but rather after it has been cut out of the patient's body by the surgeon. To do this, the piece of tissue cut away will be scanned using a specially designed PET-CT scanner.

The overall goal of this study is to gain additional knowledge. More specifically, the investigators wish to determine which medical conditions may benefit from high-resolution PET-CT specimen imaging.

DETAILED DESCRIPTION:
The rationale of this pilot study is to obtain scientific knowledge on the clinical usefulness of perioperative high-resolution PET-CT specimen imaging in different clinical indications and to document the radiation safety of perioperative high-resolution PET-CT specimen imaging.

The study will investigate the clinical value of perioperative high-resolution PET-CT specimen imaging in breast, prostate, thyroid, head & neck, skin, and primary and secondary hepatobiliary cancer, parathyroid adenoma, brain cancer, suspected malignant and benign gastrointestinal lesions, neuro-endocrine malignancies, genitourinary malignancies (including bladder cancer, renal pelvis and ureter carcinoma, adrenal cortical carcinoma and renal cell carcinoma), thoracovascular malignancies and in patients undergoing biopsy after metabolic active lesions were detected.

The secondary objectives of the study are:

* to correlate the margin status based on high-resolution PET-CT specimen images with the margin status based on microscopic histopathological analysis;
* to compare the visualization of the target lesion between perioperative high-resolution PET-CT specimen imaging and pre-operative standard-of-care imaging (e.g. whole-body PET-CT imaging, MRI imaging etc);

ELIGIBILITY:
A. Inclusion Criteria:

* able to understand treatment protocol and informed consent form
* estimated by the investigator to be compliant for study participation

  1. Fulfilling all group-specific inclusion criteria:
* confirmed breast cancer with an indication to undergo breast conserving surgery
* confirmed prostate cancer with an indication to undergo resective surgeryprostatectomy;
* confirmed thyroid lesion with an indication to undergo resective surgery;
* confirmed parathyroid adenoma with an indication to undergo resective surgery;
* suspected basal cell carcinoma, squamous cell carcinoma or melanoma with an indication to undergo resective surgery;
* suspected lesion in genitourinary sites (including bladder cancer, renal pelvis and ureter carcinoma, adrenal cortical carcinoma and renal cell carcinoma) with an indication to undergo resective surgery;
* suspected lesion in the head & neck region with an indication to undergo resective surgery;
* confirmed primary or secondary hepatobiliary cancer with an indication to undergo resective surgery;
* patients undergoing biopsy after metabolic active lesions were detected on a PET scan.
* suspected neuro-endocrine malignancies with an indication to undergo resective surgery.
* suspected brain tumor with an indication to undergo resective surgery.
* Suspected malignant and benign gastrointestinal lesions with an indication to undergo resective surgery.
* suspected malignant thoracovascular lesions with an indication to undergo resective surgery

B. Exclusion Criteria:

* general or local contra-indications for resective surgery;
* in case of FDG-based PET tracers: a blood glucose level over 200 mg/dL on the day of surgery;
* pregnancy or lactation;
* participation in other clinical studies with a radiation exposure of more than 1 mSv in the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-08-06 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of margin status | Up to 2 weeks after surgery (histopathology results)
  to correlate the margin status based on high-resolution PET-CT specimen images with the margin status based on microscopic histopathological analysis

SECONDARY OUTCOMES:
Comparison of the visualization of the target lesion | From pre-operative imaging until imaging during surgery
  post-hoc comparison of the visualization of the target lesion between perioperative high-resolution PET-CT specimen imaging and pre-operative standard-of-care imaging (if recent pre-operative scan available). This will include lesion dimensions (e.g. delineation based on percentage of SUVmax) but also tumor to background ratio variability;

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Maria Middelares, Ghent, Oost Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided